CLINICAL TRIAL: NCT03390985
Title: Canadian Observation Trial in CF Patients Undergoing Treatment With Ivacaftor
Acronym: G551D
Status: Completed | Type: Observational
Sponsor: Tanja Gonska (Other)
Responsible Party: Sponsor-Investigator, Tanja Gonska, Principal Investigator, The Hospital for Sick Children
Organization: The Hospital for Sick Children (Other)
Other Study IDs: 1000036224
Record Dates: First submitted 2017-12-18; First posted 2018-01-05 (Actual); Last update posted 2018-01-05 (Actual); Status verified 2017-12

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — sputum, stool, plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Specific aims:

1. To elucidate the biological mechanism that leads to pulmonary and nutritional improvement in CF patients following treatment with ivacaftor using advanced techniques to assess changes of the pulmonary and nutritional status
2. To examine the relation between the individual response to ivacaftor and the presence of modifier genes associated with CF disease severity,
3. To assess altered CFTR function using new available in vivo tests,
4. To validate newly developed in vivo sweat tests with well established functional tests,
5. To establish correlation between the CFTR response to Vx-770 measured in a new ex vivo method (organoids) and the actual clinical and/or functional response in individual patients,
6. To examine response in other CF-specific features such as aqua wrinkling.
7. To examine if sleep/activity level changes.
8. To establish a biorepository to enable further investigations.

ELIGIBILITY:
Inclusion Criteria:

* any patient being prescribed ivacaftor

Exclusion Criteria:

* only relates to specific tests

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: CF patients with any of the following mutations G551D, G178R, S549N, S549R, G551S, G1244E, S1251N, S1255P, G1349D and G970R approved by Health Canada to receive ivacaftor.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2013-04-23 (Actual); Primary Completion 2017-07-26 (Actual); Study Completion 2017-07-26 (Actual)

PRIMARY OUTCOMES:
Functional in vivo Cystic fibrosis transmembrane conductor regulator (CFTR) tests: Nasal Potential difference (NPD) measurements | 7 study visits over a 2 year period
  NPD is measured to assess CFTR function as difference in mV between post and pre-drug start
Functional in vivo test: Beta-adrenergic sweat secretion test | 7 study visits over a 2 year period
  The beta-adrenergic sweat secretion test is measured as ratio of beta-adrenergic/cholinergic sweat secretion as difference between post and pre-drug start
Functional in vitro test: Rectal tissue biopsies to measure CFTR function in vitro using Ussing chamber studies and organoids | one study visit
  Rectal tissue specimen is being used to measure the response to ivcaftor of individual CF patients in vitro
Functional in vitro test: Collect nasal brushes for CFTR to generate nasal cell cultures for the assessment of ivacaftor response and CFTR function | 2 study visits in 6 months
  Nasal cultures are used to measure the response to ivcaftor in vitro as difference of the forskolin-induced response of CFTR to ivacaftor

SECONDARY OUTCOMES:
Measurement of aqua wrinkling | 2 study visits in 3 months
  CF patients response to submerge in water for 5 min to develop a skin phenomenon known as aqua wrinkling is being measured subjectively pre and post-drug
Measurement of exhaled fractionated nitrogen oxide (FeNo) | 5 study visits in 1 year
  the fraction of the exhaled NO in % In the expiration of CF patients is being measured pre-and post-drug
Measurements of the lung clearance index | 5 study visits in 1 year
  Multiple breath wash-out technique is being used to measure the lung clearance index (no unit) pre and post-drug
Measurements of the pancreas function using fecal elastase test | 4 study visits in 2 years
  Fecal elastase in stool is determined in microg/g stool pre and post-drug
Measurements of the pancreas function using serum trypsinogen | 4 study visits in 2 years
  Serum trypsinogen is determined in nmol/L pre and post-drug
Assessment of the nutritional status | 4 study visits in 2 years
  Nutritional status is assessed using the BODPOD in kg fat or non-fat mass change or percentage fat or non-fat mass change pre and post-drug
Measurements of the resting energy expenditure | 4 study visits in 2 years
  The resting energy expenditure is measured using indirect calorimetry in kcal/d pre and post-post
Assessment of pulmonary radiological changes using high resolution CT | 4 study visits in 2 years
  Radiological pulmonary changes are being assessed using high resolution CT pre and post-drug (descriptive and Bhalla score)
Assessment of glucose tolerance | 4 study visits in 2 years
  Glucose tolerance is being assessed using the organ glucose tolerance test and glucose levels 2 hrs post in mmol/L will be compared pre and post-drug

IPD SHARING:
Plan to Share IPD: No